CLINICAL TRIAL: NCT01057095
Title: Mechanisms of PLAGL2-Induced Leukaemogenesis
Brief Title: Studying Gene Expression in Tissue Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B12; COG-AAML10B12 (Other: Children's Oncology Group); CDR0000664240 (Other: Clinical Trials.gov); NCI-2011-02208 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at gene expression in tissue samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Screen acute myeloid leukemia (AML) samples to correlate high relative expression levels of PLAGL2 and putative PLAGL2 target genes (implicated in microarray study) with potential pathogenic relevance with respect to AML development.

OUTLINE: Cryopreserved mRNA from diagnostic samples is analyzed for gene expression by reverse transcriptase-PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia, including inv(16)(p13;q22) abnormalities

  * No t(15;17)(q22;q12) or t(8;21)(q22;q22) abnormalities

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Correlation of high relative expression levels of PLAGL2 and putative PLAGL2 target genes with potential pathogenic relevance

CONTACTS AND LOCATIONS:
Overall Officials: Soheil Meshinchi, MD, Principal Investigator — Fred Hutchinson Cancer Center